CLINICAL TRIAL: NCT04175002
Title: Endometrial Heparin-binding Epidermal Growth Factor Expression in Implantation Window of Obese Women With Polycystic Ovarian Syndrome(PCOS)
Brief Title: Endometrial Heparin-binding Epidermal Growth Factor Expression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Azrai Abu, Principal Investigator, National University of Malaysia
Other Study IDs: UKM PPI.800-1/1/5/JEP-2019-367
Record Dates: First submitted 2019-11-18; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Gene Abnormality
Keywords: heparin-binding epidermal growth factor; polycystic ovarian syndrome; implantation window; obese
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity | interventions — Utrogestan

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — endometrial tissue, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Anovulatory PCOS women with a BMI greater than 27
  Interventions: Drug: utrogestan
- Anovulatory PCOS women with a BMI lower than 25
  Interventions: Drug: utrogestan
- Healthy fertile women with a BMI greater than 27
- Healthy fertile women with a BMI lower than 25

INTERVENTIONS:
Drug: utrogestan — oral uterogeston 200mg daily to achieve window of implantation from previous study
  Groups: Anovulatory PCOS women with a BMI greater than 27; Anovulatory PCOS women with a BMI lower than 25

SUMMARY:
Women with PCOS comprise a majority of fertility clinic attendees. Unfortunately, a high failure rate following fertility treatment was observed especially in obese women due to implantation failure. The local study on PCOS women has shown significant changes in an endometrial tumor - regulatory genes but not focusing on the endometrial implantation failure. Many previous attempts using human chorionic gonadotrophin (HCG) infused embryo, gonadotrophin agonist therapy or progesterone support aiming to improve implantation failure in the assisted reproductive technique still unable to enhance pregnancy rate beyond 40% despite a higher' fertilization rate up to 95%. There is still a research gap on what makes obese PCOS women prone to coincides with implantation failure. Endometrial component related to the expression of growth factors play an integral role in establishing cellular context necessary for successful pregnancy. Thus, a new fundamental knowledge on endometrial specific heparin-binding epidermal growth factor expression in the obese PCOS women is vitally important, not only to predict implantation failure but a potential therapy to improve pregnancy outcome.

DETAILED DESCRIPTION:
This prospective study is going to be performed at UKM Medical Centre for a duration of 1 year. The PCOS and control women will be recruited from the Medically Assisted clinic in Obstetrics & Gynaecology department.

The sample size of this study is calculated using Power and Sample Size Calculator by Dupont & Plummer 1998 for paired t-test response version 3.1.2; using the endpoint of mean of Hb-EGF expression during window of implantation in predicting successful pregnancy following in vitro fertilization (IVF) rate by Mengling et al. 2016 (11) as one of its specific outcome. The auto-generated sample size using this programme is 8 subjects. Considering the dropout rate of the sample is 30%, the total sample size required in this study is 10 subjects each arm, making a total sample size 40.

The participants are divided into four groups according to PCOS diagnosis and Asian adult population body mass index (BMI):

1. Anovulatory PCOS women with a BMI greater than 27 (OB-PCOS)
2. Anovulatory PCOS women with a BMI lower than 25 (NW-PCOS)
3. Healthy fertile women with a BMI greater than 27 (OB-C)
4. Healthy fertile women with a BMI lower than 25 (NW-C)

In the PCOS group, generally anovulatory cycle hence the implantation window during mid-secretory endometrium can be exhibit following a daily oral micronized progesterone (Utrogestan 200mg) for 10 days based on previously published methods.

Volunteers in the control group with a normal regular menses will be counseled regarding the procedure and monitored for ovulation. The endometrial biopsy will be acquired during implantation window (mid-secretory endometrium), which occurred 7-9 days after the ultrasound and urinary LH confirmed ovulation.

Endometrial samples are obtained using the Pipelle de Cornier catheter for all participants. The endometrium sample that is taken is divided into two portions; a portion for histopathological examination (HPE) for endometrial dating and a portion frozen in liquid nitrogen at -80 degrees Celsius for real-time PCR analysis.

For endometrial dating, all samples were analyzed by classical histological analysis according to the criteria of Noyes.

A total amount of RNA was isolated from the endometrial tissue using RNA easy kit by following manufacturer's instruction. Pellet will be suspended in 30ul of RNAase-DNAse free water. Finally, nanodrop will be used to determine the concentration and quality of RNA. By following manufacture's instruction, total RNA will be reversed transcribed to cDNA. The target for cDNA is primers for heparin binding epidermal growth factor. QRT-PCR will be performed using Sybergreen Master Mix and detected using QRT-PCR detector machine in accordance with manufacturer's protocols. The reaction was running in real-time PCR machine with 40 cycles and cycling temperature as follows: 95 ºC for 10 minutes and 15 seconds, 56 ºC for 30 seconds and final dissociation stage: 94 ºC for 15 seconds, 56 ºC for 15 seconds and last 95 ºC for 15 seconds. Relative quantification will be calculated by normalizing against any housekeeping genes available. Positive controls and negative controls will be included in each analysis run.

ELIGIBILITY:
The inclusion criteria for the study group are:

1. All patients between the aged of 18 to 40 years.
2. Women diagnosed with polycystic ovarian syndrome fulfilling two out of three Rotterdam criteria (ie, oligo- or anovulation, hyperandrogenism, and polycystic ovaries on ultrasound).
3. Healthy volunteer with confirmed fertility (having at least one child previously), with a normal level of basic reproductive hormones and regular interval of the menstrual cycle (26 to 32 days). (Control group)

The exclusion criteria are:

1. Smoking
2. any hormonal treatment or other drugs to treat anovulation for at least 3 months before the study
3. Pregnancy or lactation during the preceding 12 months
4. Systemic disease such as endocrine or eating disorders besides PCOS
5. Diagnosed with a uterine or ovarian disease.
6. Any regular medication such as hormones, herbal substance, statins or corticoids for at least 3 months before the study.
7. History of intrauterine device placement.

The inclusion criteria for the control group are:

1. All patients between the aged of 18 to 40 years.
2. Healthy volunteer with confirmed fertility (having at least one child previously), with a normal level of basic reproductive hormones and regular interval of the menstrual cycle (26 to 32 days).

The exclusion criteria are:

1. Smoking
2. any hormonal treatment or other drugs to treat anovulation for at least 3 months before the study
3. Pregnancy or lactation during the preceding 12 months
4. Systemic disease such as endocrine or eating disorders besides PCOS
5. Diagnosed with a uterine or ovarian disease.
6. Any regular medication such as hormones, herbal substance, statins or corticoids for at least 3 months before the study.
7. History of intrauterine device placement.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This prospective study is going to be performed at UKM Medical Centre for a duration of 1 years. The PCOS and control women will be recruited from the Medically Assisted clinic in Obstetrics & Gynaecology department.
  Patients will be recruited following written consent. Background information such as age, race, parity, menstrual pattern, associated symptoms will be taken. Clinical assessment which includes height, weight, body mass index and hirsutism (determined by a modified Ferriman and Gallwey score) will be performed. The serum levels of follicle-stimulating hormone (FSH), luteinizing hormone (LH), total testosterone (TT), cortisol, prolactin (PRL), dehydroepiandrosterone sulfate (DHEAS), and β-human chorionic gonadotropin (β-hCG) are measured for all participants. A transvaginal ultrasound scan of the ovaries will be obtained. Endometrial samples are obtained using the Pipelle de Cornier catheter for all participant
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Endometrial Heparin-binding Epidermal Growth Factor Expression | After 10 days of oral uterogeston 20mg daily
  For obese and normal BMI PCOS window of implantation based on Noyes criteria
Endometrial Heparin-binding Epidermal Growth Factor Expression | After 5 days of positive urinary LH
  For obese and normal BMI normal fertile women window of implantation based on Noyes criteria

SECONDARY OUTCOMES:
Hormonal assay | During day 2-6 of menstrual cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Medically Assisted clinic in Obstetrics & Gynaecology department, UKM Medical Centre, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mengling S, Xian X, Yongli L, et al. Expression of heparin-binding epidermal growth factor in the endometrium is positively correlated with IVF-ET pregnancy outcome. Int J Clin Exp Pathol 2016;9(8):8280-8285.
- [Result] Fauser BC, Tarlatzis BC, Rebar RW, Legro RS, Balen AH, Lobo R, Carmina E, Chang J, Yildiz BO, Laven JS, Boivin J, Petraglia F, Wijeyeratne CN, Norman RJ, Dunaif A, Franks S, Wild RA, Dumesic D, Barnhart K. Consensus on women's health aspects of polycystic ovary syndrome (PCOS): the Amsterdam ESHRE/ASRM-Sponsored 3rd PCOS Consensus Workshop Group. Fertil Steril. 2012 Jan;97(1):28-38.e25. doi: 10.1016/j.fertnstert.2011.09.024. Epub 2011 Dec 6. PMID 22153789
- [Result] Joham AE, Boyle JA, Ranasinha S, Zoungas S, Teede HJ. Contraception use and pregnancy outcomes in women with polycystic ovary syndrome: data from the Australian Longitudinal Study on Women's Health. Hum Reprod. 2014 Apr;29(4):802-8. doi: 10.1093/humrep/deu020. Epub 2014 Feb 18. PMID 24549213
- [Result] Bellver J, Martinez-Conejero JA, Labarta E, Alama P, Melo MA, Remohi J, Pellicer A, Horcajadas JA. Endometrial gene expression in the window of implantation is altered in obese women especially in association with polycystic ovary syndrome. Fertil Steril. 2011 Jun;95(7):2335-41, 2341.e1-8. doi: 10.1016/j.fertnstert.2011.03.021. Epub 2011 Apr 9. PMID 21481376
- [Result] Schulte MM, Tsai JH, Moley KH. Obesity and PCOS: the effect of metabolic derangements on endometrial receptivity at the time of implantation. Reprod Sci. 2015 Jan;22(1):6-14. doi: 10.1177/1933719114561552. Epub 2014 Dec 7. PMID 25488942
- [Result] DeUgarte DA, DeUgarte CM, Sahakian V. Surrogate obesity negatively impacts pregnancy rates in third-party reproduction. Fertil Steril. 2010 Feb;93(3):1008-10. doi: 10.1016/j.fertnstert.2009.07.1005. Epub 2009 Sep 5. PMID 19733847
- [Result] Piltonen TT. Polycystic ovary syndrome: Endometrial markers. Best Pract Res Clin Obstet Gynaecol. 2016 Nov;37:66-79. doi: 10.1016/j.bpobgyn.2016.03.008. Epub 2016 Apr 1. PMID 27156350
- [Result] Large MJ, Wetendorf M, Lanz RB, Hartig SM, Creighton CJ, Mancini MA, Kovanci E, Lee KF, Threadgill DW, Lydon JP, Jeong JW, DeMayo FJ. The epidermal growth factor receptor critically regulates endometrial function during early pregnancy. PLoS Genet. 2014 Jun 19;10(6):e1004451. doi: 10.1371/journal.pgen.1004451. eCollection 2014 Jun. PMID 24945252
- [Result] Lim HJ, Dey SK. HB-EGF: a unique mediator of embryo-uterine interactions during implantation. Exp Cell Res. 2009 Feb 15;315(4):619-26. doi: 10.1016/j.yexcr.2008.07.025. Epub 2008 Aug 3. PMID 18708050
- [Result] Jessmon P, Leach RE, Armant DR. Diverse functions of HBEGF during pregnancy. Mol Reprod Dev. 2009 Dec;76(12):1116-27. doi: 10.1002/mrd.21066. PMID 19565643
- [Result] Wirstlein PK, Mikolajczyk M, Skrzypczak J. Correlation of the expression of heparanase and heparin-binding EGF-like growth factor in the implantation window of nonconceptual cycle endometrium. Folia Histochem Cytobiol. 2013;51(2):127-34. doi: 10.5603/FHC.2013.0020. PMID 23907942
- [Result] Zang H, Sahlin L, Masironi B, Eriksson E, Linden Hirschberg A. Effects of testosterone treatment on endometrial proliferation in postmenopausal women. J Clin Endocrinol Metab. 2007 Jun;92(6):2169-75. doi: 10.1210/jc.2006-2171. Epub 2007 Mar 6. PMID 17341565
- [Result] Hulchiy M, Nybacka A, Sahlin L, Hirschberg AL. Endometrial Expression of Estrogen Receptors and the Androgen Receptor in Women With Polycystic Ovary Syndrome: A Lifestyle Intervention Study. J Clin Endocrinol Metab. 2016 Feb;101(2):561-71. doi: 10.1210/jc.2015-3803. Epub 2015 Dec 9. PMID 26649621
- [Result] Apparao KB, Lovely LP, Gui Y, Lininger RA, Lessey BA. Elevated endometrial androgen receptor expression in women with polycystic ovarian syndrome. Biol Reprod. 2002 Feb;66(2):297-304. doi: 10.1095/biolreprod66.2.297. PMID 11804942
- [Derived] Hamid FA, Mokhtar MH, Abdul Karim AK, Ahmad MF, Abd Aziz NH, Abdul Wahab AY, Abu MA. Obesity results in lower integrin expression in women with polycystic ovarian syndrome during the window of implantation. Front Endocrinol (Lausanne). 2025 Oct 21;16:1590716. doi: 10.3389/fendo.2025.1590716. eCollection 2025. PMID 41195204